CLINICAL TRIAL: NCT03024684
Title: Statin for Preventing Hepatocellular Carcinoma Recurrence After Curative Treatment: a Double-blind Randomized Placebo-controlled Trial
Brief Title: Statin for Preventing Hepatocellular Carcinoma Recurrence After Curative Treatment
Acronym: SHOT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Collaborators: E-DA Hospital (Other); National Taiwan University Hospital (Other); Taichung Veterans General Hospital (Other); Mackay Memorial Hospital (Other); Tainan Municipal Hospital (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 105005
Record Dates: First submitted 2017-01-15; First posted 2017-01-19 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: HepatoCellular Carcinoma
Keywords: Hepatocellular carcinoma; statin; curative ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin (Experimental): Atorvastatin 10mg oral once daily
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Matched placebo (sugar pill) once daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10mg daily
  Arms: Statin
Drug: Placebo Oral Tablet — Placebo one tablet daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether statin could prevent recurrence of hepatocellular carcinoma after curative treatment

DETAILED DESCRIPTION:
This is a multi-center double-blind randomized placebo-controlled trial. A total of 240 patients with HCC at BCLC stage 0 or A will be enrolled from 8 hospitals in Taiwan. After complete ablation or hepatic resection of the tumor(s), participants are randomized 1:1 to receive either atorvastatin 10mg once daily (intervention group) or matched placebo (control group) for 3 years. During the 3-year period, patients are monitored for recurrence of HCC by dynamic computed tomography (or magnetic resonance image) every 4 months. They will be followed up until death, withdrawal from participation, study termination, or 3 years after the ablative treatment. The primary endpoint is to compare the 3-year cumulative incidence of recurrent HCC between the intervention group and control counterpart. Secondary endpoints are occurrence of clinical complications related to hepatic decompensation (including gastroesophageal variceal bleeding, spontaneous peritonitis, hepatic encephalopathy, hepatorenal syndrome, and hepatopulmonary syndrome), liver-related mortality, and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with HCC BCLC stage 0 or A who received curative radiofrequency ablation or hepatic resection could be eligible.
* Individuals who had single HCC (size > 5.0 cm) received hepatic resection would be eligible
* Individuals with prior history of HCC who had ever received curative ablation or hepatic resection without any recurrence for more than 2 years could be eligible if they had a new episode of recurrent HCC which could meet either of the former two criteria.
* After 12+/-1 weeks of curative treatment, eligible patients who have no evidence of local residual or recurrent tumors according to the dynamic CT or MRI could be enrolled
* The diagnosis of fresh HCC should be compatible with either pathological report or meet the criteria of AASLD guidelines

Exclusion Criteria:

* Undetermined nature of hepatic tumor
* HCC with extrahepatic metastasis or major vascular invasion
* With other malignant disease
* Child Pugh score >7
* Previous history of CAD event (angina, unstable angina, acute myocardial infarction) or ischemic stroke
* Hyperlipidemia or other indication for statin (according to Taiwan NHI guideline)
* Advanced CKD (eGFR<30) or ESRD
* Severe comorbidity with life expectancy < 2 years
* Allergy to statin

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
3-year cumulative incidence of recurrent HCC between the intervention group and control counterpart | 3 years
  Recurrence rate of HCC

SECONDARY OUTCOMES:
occurrence of clinical complications related to hepatic decompensation | 3 years
  clinical complications or hepatic decompensation

CONTACTS AND LOCATIONS:
Overall Officials: Po Yueh Chen, Doctor, Principal Investigator — Ditmanson Medical Foundation Chia-Yi Christian Hospital
Locations (6):
- Taiwan (6):
  - Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City
  - E-DA Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Tainan Municipal Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital Yun-Lin Branch, Yunlin

IPD SHARING:
Plan to Share IPD: No